CLINICAL TRIAL: NCT00771862
Title: Prevention of Phantom Limb and Stump Pain Using Ambulatory Continuous Peripheral Nerve Blocks: A Pilot Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Could not secure funding to complete the study.
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Phantom Pain Prevention PILOT
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Amputation; Phantom Limb Pain; Stump Pain
Keywords: pain; amputation; phantom limb; stump pain; catheter; nerve block; peripheral nerve block; ucsd; post-amputation phantom limb or stump pain
MeSH Terms: conditions — Phantom Limb; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. standard care (Placebo Comparator): 1 day of perineural ropivacaine 0.2% infusion followed by 4-5 days of normal saline infusion.
  Interventions: Procedure: perineural ropivicaine
- 2: experimental care (Active Comparator): 4-5 days of perineural ropivacaine 0.4% infusion.
  Interventions: Procedure: perineural ropivicaine

INTERVENTIONS:
Procedure: perineural ropivicaine — Subjects will be randomized to one of two groups: ropivicaine 0.2% infusion for days 0-1 then infusion with normal saline (placebo) for days 1 through catheter removal (POD 4 or 5) or ropivicaine 0.4% infusion for day 0 through catheter removal (POD 4 or 5). The infusion rate will be set at 7-11 mL/h.

SUMMARY:
The purpose of this research study is to determine if putting local anesthetic through one or two percutaneous catheters placed next to the nerves that go to an amputated limb will decrease long-term pain in the amputated limb.

DETAILED DESCRIPTION:
Specific Aim 1: To determine if, compared with current and customary analgesia, the addition of multiple-day ambulatory continuous peripheral nerve blocks decrease the incidence and severity of post-amputation phantom limb and stump pain.

Hypothesis 1: Following upper or lower extremity amputation, the incidence of phantom limb and/or stump pain will be significantly decreased four weeks following multiple-day ambulatory continuous peripheral nerve blocks as compared with patients receiving standard-of-care treatment.

Hypothesis 2: Following upper or lower extremity amputation, the severity of phantom limb and/or stump pain will be significantly decreased four weeks following multiple-day ambulatory continuous peripheral nerve blocks as compared with patients receiving standard-of-care treatment (as measured on the 11-point numeric rating scale).

ELIGIBILITY:
Inclusion Criteria:

* undergoing unilateral surgical amputation of the upper or lower extremity including at least one metacarpal or metatarsal bone, respectively
* currently without phantom limb and/or stump pain in a previously-amputated limb
* ages 18 years or older
* desiring perineural infusion for up to 6 days
* willing to have an ambulatory infusion following hospital discharge

Exclusion Criteria:

* hepatic or renal failure
* allergy to the study medications
* pregnancy
* incarceration
* possessing a contraindication to perineural catheter placement or perineural local anesthetic infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome measurement will be the difference in average NRS (as administered as part of the Brief Pain Inventory) at 4 weeks between the two treatment groups. | Week 4

SECONDARY OUTCOMES:
Pain and Physical functioning: Brief Pain Inventory (includes the 11-point numeric rating scale of pain intensity) | Preoperative, then days 3, 8, 28, 84, and 365
Emotional Functioning: Beck Depression Inventory | Preoperative, then days 28 and 365
The incidence of phantom limb and/or stump pain will be significantly decreased four weeks following multiple-day ambulatory continuous peripheral nerve blocks as compared with patients receiving standard-of-care treatment. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States